CLINICAL TRIAL: NCT05738850
Title: Generalized Anxiety Disorder (GAD): A First-in-Human Single Ascending Dose and Food Effect Study of ABBV-932 in Healthy Adult Subjects
Brief Title: Study to Assess Adverse Events and How ABBV-932 Oral Capsules Moves Through the Body of Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Gedeon Richter Plc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M23-889
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Generalized Anxiety Disorder (GAD); Healthy Participants
Keywords: Generalized Anxiety Disorder (GAD); ABBV-932
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- Part 1: ABBV-932 (Experimental): Participants will receive ABBV-932 on Day 1 and followed for 30 days.
  Interventions: Drug: ABBV-932
- Part 1: Placebo (Placebo Comparator): Participants will receive placebo on Day 1 and followed for 30 days.
  Interventions: Drug: Placebo
- Part 2: Sequence 1 (Experimental): Participants will receive ABBV-932 on Day 1 in Period 1 under fasting conditions and followed for 30 days. Participants will receive ABBV-932 with food on Day 1 in Period 2 and followed for 30 days.
  Interventions: Drug: ABBV-932
- Part 2: Sequence 2 (Experimental): Participants will receive ABBV-932 with food on Day 1 in Period 1 and followed for 30 days. Participants will receive ABBV-932 on Day 1 in Period 2 under fasting conditions and followed for 30 days.
  Interventions: Drug: ABBV-932
- Part 3: Japanese Participants: ABBV-932 (Experimental): Japanese participants will receive ABBV-932 on Day 1 in Period 1 and followed for 30 days.
  Interventions: Drug: ABBV-932
- Part 3: Japanese Participants: Placebo (Placebo Comparator): Japanese participants will receive placebo on Day 1 in Period 1 and followed for 30 days.
  Interventions: Drug: Placebo
- Part 3: Han-Chinese Participants: ABBV-932 (Experimental): Han-Chinese participants will receive placebo on Day 1 in Period 1 and followed for 30 days.
  Interventions: Drug: ABBV-932

INTERVENTIONS:
Drug: ABBV-932 — Oral Capsule
  Arms: Part 1: ABBV-932; Part 2: Sequence 1; Part 2: Sequence 2; Part 3: Han-Chinese Participants: ABBV-932; Part 3: Japanese Participants: ABBV-932
Drug: Placebo — Oral Capsule
  Arms: Part 1: Placebo; Part 3: Japanese Participants: Placebo

SUMMARY:
The main objective of this study is to assess pharmacokinetics, safety, and tolerability of ABBV-932 in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Parts 1 and 2: Healthy individuals with body-mass index (BMI) >= 18.0 to <= 32.0 kg/m2, rounded to the tenths decimal.
* Part 3: Healthy Japanese, Han Chinese individuals with BMI >= 18.0 to <= 30.0 kg/m2, rounded to the tenths decimal.
* Condition of general good health based upon the results of a medical history, physical examination, vital signs, laboratory profile, neurological examination, and a 12-lead ECG.

Exclusion Criteria:

- History of any clinically significant illness/infection/major febrile illness, hospitalization, or any surgical procedure within 30 days prior to the first dose of study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of ABBV-932 | Up to approximately 5 days
  Cmax of ABBV-932.
Time to Cmax (Tmax) of ABBV-932 | Up to approximately 5 days
  Tmax of ABBV-932.
Terminal Phase Elimination Rate Constant (Beta) of ABBV-932 | Up to approximately 5 days
  Terminal phase elimination rate constant (beta) of ABBV-932.
Terminal Phase Elimination Half-Life (t1/2) of ABBV-932 | Up to approximately 5 days
  Terminal phase elimination half-life of ABBV-932.
Area Under the Concentration-Time Curve From Time 0 to Time t (AUCt) of ABBV-932 | Up to approximately 5 days
  AUCt of ABBV-932.
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of ABBV-932 | Up to approximately 5 days
  AUCinf of ABBV-932.
Maximum Plasma Concentration (Cmax) of DCAR | Up to approximately 5 days
  Cmax of DCAR.
Time to Cmax (Tmax) of DCAR | Up to approximately 5 days
  Tmax of DCAR.
Terminal Phase Elimination Rate Constant (Beta) of DCAR | Up to approximately 5 days
  Terminal phase elimination rate constant (beta) of DCAR.
Terminal Phase Elimination Half-Life (t1/2) of DCAR | Up to approximately 5 days
  Terminal phase elimination half-life of DCAR.
Area Under the Concentration-Time Curve From Time 0 to Time t (AUCt) of DCAR | Up to approximately 5 days
  AUCt of DCAR.
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of DCAR | Up to approximately 5 days
  AUCinf of DCAR.
Maximum Plasma Concentration (Cmax) of DDCAR | Up to approximately 5 days
  Cmax of DDCAR.
Time to Cmax (Tmax) of DDCAR | Up to approximately 5 days
  Tmax of DDCAR.
Terminal Phase Elimination Rate Constant (Beta) of DDCAR | Up to approximately 5 days
  Terminal phase elimination rate constant (beta) of DDCAR.
Terminal Phase Elimination Half-Life (t1/2) of DDCAR | Up to approximately 5 days
  Terminal phase elimination half-life of DDCAR.
Area Under the Concentration-Time Curve From Time 0 to Time t (AUCt) of DDCAR | Up to approximately 5 days
  AUCt of DDCAR.
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of DDCAR | Up to approximately 5 days
  AUCinf of DDCAR.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (2):
- United States (2):
  - Anaheim Clinical Trials LLC /ID# 254178, Anaheim, California
  - Acpru /Id# 249639, Grayslake, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-889